CLINICAL TRIAL: NCT00167258
Title: Effectiveness and Costs of Enhanced Cocaine Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Dr. James McKay, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 702110
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

INTERVENTIONS:
Behavioral: Voucher Reinforcement
Behavioral: Extra Counseling Services
Behavioral: Voucher Reinforcement + Extra Counseling Services

SUMMARY:
The study will evaluate the effectiveness, economic benefits, and costs of voucher reinforcement for cocaine and alcohol abstinence, additional counseling services, and their combination in a sample of cocaine dependent patients receiving outpatient treatment as usual in a community clinic.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in an intensive outpatient program (IOP) for no more than 1 month
* Current DSM-IV diagnosis of cocaine dependence (month prior to IOP treatment)
* 18-65 years of age
* Ability to provide names of informants to help locate subject for follow-up

Exclusion Criteria:

* IV heroin use in last year
* Acute medical/psychiatric diagnosis that precludes outpatient treatment
* Inpatient treatment for 6 weeks or more prior to IOP treatment
* Incarceration for 6 months or more prior to IOP treatment

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: James R McKay, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States